CLINICAL TRIAL: NCT06025474
Title: Comparative Evaluation of Vortioxetine Versus Other Antidepressants With Pregabalin Augmentation in Treatment-resistant Burning Mouth Syndrome: a Prospective Longitudinal Clinical Trial With Treatment Response Prediction
Brief Title: Comparison of Vortioxetine Versus Other Antidepressants With Pregabalin Augmentation in Burning Mouth Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Daniela Adamo, Clinical Assistant, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 251/19
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Burning Mouth Syndrome
Keywords: Burning mouth syndrome; vortioxetine; pregabalin; Drug Therapy
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Vortioxetine; Paroxetine; Tablets; Sertraline; Citalopram; Escitalopram; Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Vortioxetine+Pregabalin (Experimental): VO group(20mg)+ PGB (75mg) N= 136 Vortioxetine 20 mg, encapsulated tablets, orally, once daily, then pregabalin 75 mg, encapsulated tablets, orally, once daily. Pregabalin (75mg/day) was added, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks
  Interventions: Drug: Vortioxetine 20Mg Tab; Drug: Pregabalin 75mg
- Paroxetine+Pregabalin (Active Comparator): P group (20mg) + PGB (75mg); N= 10 Paroxetine 20 mg, encapsulated tablets, orally, once daily, then pregabalin 75 mg, encapsulated tablets, orally, once daily. Pregabalin (75mg/day) was added, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks
  Interventions: Drug: Paroxetine 20 Mg Oral Tablet; Drug: Pregabalin 75mg
- Sertraline+Pregabalin (Active Comparator): S group (50mg) + PGB (75mg); N= 8 Sertraline 50 mg, encapsulated tablets, orally, once daily, then pregabalin 75 mg, encapsulated tablets, orally, once daily. Pregabalin (75mg/day) was added, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks
  Interventions: Drug: Sertraline 50 MG; Drug: Pregabalin 75mg
- Citalopram+Pregabalin (Active Comparator): C group (20mg)+ PGB (75mg) N= 8 Citalopram 20 mg, encapsulated tablets, orally, once daily, then pregabalin 75 mg, encapsulated tablets, orally, once daily. Pregabalin (75mg/day) was added, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks
  Interventions: Drug: Citalopram 20mg; Drug: Pregabalin 75mg
- Escitalopram+Pregabalin (Active Comparator): E group (10mg) + PGB (75mg); N= 8 Escitalopram 10 mg, encapsulated tablets, orally, once daily, then pregabalin 75 mg, encapsulated tablets, orally, once daily. Pregabalin (75mg/day) was added, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks
  Interventions: Drug: Escitalopram 10mg; Drug: Pregabalin 75mg
- Duloxetine+Pregabalin (Active Comparator): D group (60mg)+ PGB (75mg) N= 33 Duloxetine 60 mg, encapsulated tablets, orally, once daily, then pregabalin 75 mg, encapsulated tablets, orally, once daily. Pregabalin (75mg/day) was added, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks
  Interventions: Drug: Duloxetine 60 MG; Drug: Pregabalin 75mg

INTERVENTIONS:
Drug: Vortioxetine 20Mg Tab — Encapsulated vortioxetine immediate release tablets, once daily
  Other Names: Brintellix
  Arms: Vortioxetine+Pregabalin
Drug: Paroxetine 20 Mg Oral Tablet — Encapsulated paroxetine tablets, once daily
  Arms: Paroxetine+Pregabalin
Drug: Sertraline 50 MG — Encapsulated sertraline tablets, once daily
  Arms: Sertraline+Pregabalin
Drug: Citalopram 20mg — Encapsulated citalopram tablets, once daily
  Arms: Citalopram+Pregabalin
Drug: Escitalopram 10mg — Encapsulated escitalopram tablets, once daily
  Arms: Escitalopram+Pregabalin
Drug: Duloxetine 60 MG — Encapsulated duloxetine tablets, once daily
  Arms: Duloxetine+Pregabalin
Drug: Pregabalin 75mg — Encapsulated pregabalin tablets, once daily

SUMMARY:
Background: The treatment of Burning Mouth Syndrome (BMS) presents a challenge in tailoring appropriate medication for individual patients. Antidepressants have demonstrated efficacy in alleviating symptoms in most cases; however, a subset of patients exhibit limited or no response to these treatments. The augmentation with pregabalin to conventional treatment has shown promising outcomes in relieving pain and improving quality of life in chronic pain conditions. This study aimed to compare the efficacy of vortioxetine with other antidepressants (SSRIs/SNRIs) in combination with pregabalin in a cohort of unresponsive BMS patients and to predict treatment response using clinical data.

Methods: A 52-week randomized, open-label, active-controlled study was conducted, enrolling 203 BMS patients previously treated with one antidepressant for 12 weeks and non-responder to the treatment. The study sample have included two groups: Group A (136) received vortioxetine, while Group B (67) received SSRIs/SNRIs. Pregabalin (75mg/day) was added to both groups, with a potential dosage increase to 150mg/day for inadequate responders after 12 weeks.

Treatment response was assessed by measuring reduction in VAS and SF-MPQ scores (>50 or 1-2) and HAM-A and HAM-D scores (>50% or ≤7) at 12, 24, 36 and 52 weeks. Classical logistic regression with a stepwise algorithm and Random Forest machine learning models were used to predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

* patients with a confirmed diagnosis of BMS based on the International Classification of Orofacial Pain, 1st edition [International Classification of Orofacial Pain, 1st edition (ICOP) Cephalalgia, 2020]
* patients of any race or gender; complaining of oral burning recurring daily for >2 h per day for >3 months;
* normal blood test findings (including blood count, blood glucose levels, glycated hemoglobin, serum iron, ferritin and transferrin).
* BMS patients previously treated with one antidepressant for 12 weeks and non-responder to the treatment

Exclusion Criteria:

* the presence of any disease that could be recognized as a causative factor of BMS,
* a history of a psychiatric disorder or a neurological or organic brain disorder,
* a history of alcohol or substance abuse,
* the presence of Obstructive Sleep Apnea Syndrome (OSAS)
* uncontrolled hypertension, diabetes, HIV, narrow-angle glaucoma, or participants enrolled in other investigational studies.
* participants requiring continued treatment with medications that adversely interact with the study medications (eg, quinolone antibiotics, warfarin, agents inhibiting serotonin reuptake) or with hereditary problems of fructose intolerance, glucose galactose malabsorption, or sucrose isomaltase insufficiency
* pregnancy and lactation were exclusion criteria, and women of childbearing potential were required to receive a highly effective form of contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-07-24 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 times evaluation: time 0: 0 week; time 1: 12 weeks; time 2: 24 weeks; time 3: 36 weeks; time 4: 52 weeks
  The Visual Analog Scale (VAS) (Hayes and Patterson, 1921) is a well-validated unidimensional instrument for the measure of pain intensity (Hawker et al., 2011). The score is determined by measuring the distance on the line between the "no pain" and the mark of a patient mark, providing a range of scores from 0 to 10 (0 = no oral symptoms and 10 = the worst imaginable discomfort).
Short-form McGill Pain Questionnaire (SF-MPQ) | 4 times evaluation: time 0: 0 week; time 1: 12 weeks; time 2: 24 weeks; time 3: 36 weeks; time 4: 52 weeks
  the short form of the McGill Pain Questionnaire (SF-MPQ) is a measure of the quality of pain and is a multidimensional pain questionnaire, which measures the sensory, affective, and evaluative aspects of the perceived pain (Hawker et al., 2011). It comprises 15 items from the original MPQ, each scored from 0 (none) to 3 (severe). The SF-MPQ score is obtained by summing the item scores (range 0-45). There are no established critical cutoff points for the interpretation of the scores and, as for the MPQ, a higher score indicates the worse pain.

SECONDARY OUTCOMES:
Hamilton rating scale for Depression (HAM-D) | 4 times evaluation: time 0: 0 week; time 1: 12 weeks; time 2: 24 weeks; time 3: 36 weeks; time 4: 52 weeks
  The HAM-D is a clinician-administered depression assessment scale; it contains 21 items pertaining to the affective field. The scores can range from 0 to 54. A score > 7 indicates an impairment. The scores in the range of 7-17 indicate a mild depression, the scores between 18 and 24 indicate a moderate depression, and the scores >24 indicate a severe depression
Hamilton rating scale for Anxiety (HAM-A) | 4 times evaluation: time 0: 0 week; time 1: 12 weeks; time 2: 24 weeks; time 3: 36 weeks; time 4: 52 weeks
  The HAM-A (Hamilton, 1959) is a clinician-administered anxiety assessment scale. It comprises 14 items to measure both psychic anxiety and somatic anxiety. Each item is scored on a scale of 0-4, a total score <17 indicates a mild severity, 18-24 mild to moderate, and 25-30 moderate to severe (Hamilton, 1967).
Pittsburgh Sleep Quality Index (PSQI) | 4 times evaluation: time 0: 0 week; time 1: 12 weeks; time 2: 24 weeks; time 3: 36 weeks; time 4: 52 weeks
  The PSQI (Buysse et al., 1989) explores the quality of sleep over a 1-month time interval generating seven "component" scores (0-3): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction (Carpenter and Andrykowski, 1998). The total score is obtained by the sum of all the sub-scores and ranges between 0 and 21. A total score greater than five discriminates poor sleepers from good sleepers with a high sensitivity (90%-99%) and specificity (84%-87%) (Curcio et al., 2013).

OTHER OUTCOMES:
Clinical Global Impression Scale - Improvement (CGI-I) and Severity (CGI-S) | 3 times evaluation: time 1: 12 weeks; time 2: 24 weeks; time 3: 36 weeks; time 4: 52 weeks
  CGI-I scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. Clinical Global Impression Scale-Severity of Illness (CGI-S) score-by-week as fixed effects.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Napoli, Italia, Italy

REFERENCES:
- [Background] Adamo D, Calabria E, Coppola N, Pecoraro G, Mignogna MD. Vortioxetine as a new frontier in the treatment of chronic neuropathic pain: a review and update. Ther Adv Psychopharmacol. 2021 Sep 3;11:20451253211034320. doi: 10.1177/20451253211034320. eCollection 2021. PMID 34497709
- [Background] Adamo D, Pecoraro G, Coppola N, Calabria E, Aria M, Mignogna M. Vortioxetine versus other antidepressants in the treatment of burning mouth syndrome: An open-label randomized trial. Oral Dis. 2021 May;27(4):1022-1041. doi: 10.1111/odi.13602. Epub 2020 Sep 15. PMID 32790904
- [Derived] Adamo D, Canfora F, Pecoraro G, Leuci S, Coppola N, Marenzi G, Ottaviani G, Rupel K, Pellegrini L, Aria M, D'Aniello L, Mignogna MD, Albert U. Vortioxetine versus SSRI/SNRI with Pregabalin Augmentation in Treatment-Resistant Burning Mouth Syndrome: A Prospective Clinical Trial. Curr Neuropharmacol. 2025;23(7):800-819. doi: 10.2174/1570159X22999240729103717. PMID 40016875